CLINICAL TRIAL: NCT05205343
Title: Trans-Pacific Multicenter Collaborative Study of Minimally Invasive Proximal Versus Total Gastrectomy for Proximal Gastric and Gastroesophageal Junction Cancers
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0914; NCI-2022-00267 (Other: NCI-CTRP Clinical Trial Registry)
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Gastrostomy; Gastric; GastroEsophageal Cancer
MeSH Terms: interventions — Standard of Care; Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of Care: questionnaire within 30 days before your surgery and then at 1, 3, 6, and 12 months after surgery.
  The questionnaire will ask about your health, appetite, and quality of life. It should take about 3-5 minutes to complete.
  Interventions: Other: Standard of Care
- Control group: questionnaire within 30 days before your surgery and then at 1, 3, 6, and 12 months after surgery.
  The questionnaire will ask about your health, appetite, and quality of life. It should take about 3-5 minutes to complete.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Standard of Care — complete a questionnaire within 30 days before your surgery and then at 1, 3, 6, and 12 months after surgery
  Groups: Standard of Care
Other: Control Group — complete a questionnaire within 30 days before your surgery and then at 1, 3, 6, and 12 months after surgery
  Groups: Control group

SUMMARY:
To compare the symptoms of patients who have a MIPG to the symptoms of patients who have a MITG.

DETAILED DESCRIPTION:
Primary Objective:

Delineate the short-term appetite of patients who undergo minimally-invasive proximal gastrectomy (MIPG) and compare them with those of patients with gastric and gastroesophageal adenocarcinoma who undergo total gastrectomy (MITG). We hypothesize that MIPG is associated with better postoperative appetite levels compared to MITG, which would result in improved nutritional status and maintained body weight after surgery.

Secondary Objective:

- Assess patient-reported outcomes (PROs) and nutrition measures. We will use the MD Anderson Symptom Inventory Gastrointestinal Cancer Module (MDASI-GI) questionnaire with additional three experimental question items ("PRO questionnaire") to collect preoperative and postoperative patient-reported outcomes (PROs) of QoL and check fasting ghrelin levels to correlate them with reported appetite levels. We will also retrospectively investigate factors associated with improved QoL after surgery, safety of MIPG and MITG, and oncological outcomes after MIPG and MITG.

ELIGIBILITY:
Inclusion:

1. Able to speak and read English, Spanish, Japanese or Korean
2. Participants with a biopsy-confirmed diagnosis of non-metastatic gastric or GEJ adenocarcinoma, who are scheduled to undergo MIPG or MITG for curative-intention
3. Age ≥ 18

Exclusion:

1. Participants with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract
2. Participants with known narcotic dependence, with average daily dose > 5 mg oral morphine equivalent
3. Participants deemed unable to comply with study and/or follow-up procedures, at investigators' discretion
4. Participants who are pregnant (since are excluded from receiving standard-of-care MIPG or MITG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
(MDASI-GI) MD Anderson Symptom Inventory Questionnaire | 3 months after surgery
  Appetite level (reported on a 0-10 scale, in Q8 of MDASI-GI) scale 0-not present-10 as bad as you can image

CONTACTS AND LOCATIONS:
Overall Officials: Naruhiko Ikoma, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - M D Anderson Cancer Center, Houston, Texas
- Keio University School of Medicine, Tokyo, Japan
- Yonsei University College of Medicine, Soeul, South Korea

REFERENCES:
- [Derived] Ikoma N, Grotz T, Kawakubo H, Kim HI, Matsuda S, Okui J, Tomita K, Hirata Y, Nakao A, Williams LA, Wang XS, Wang X, Mansfield PF, Hyung WJ, Badgwell BD, Strong VE, Kitagawa Y. Transpacific multicenter collaborative study of minimally invasive proximal gastrectomy vs. minimally invasive total gastrectomy for proximal gastric and gastroesophageal junction cancers: 3-month follow-up results. Surg Endosc. 2025 Dec;39(12):8371-8384. doi: 10.1007/s00464-025-12257-4. Epub 2025 Sep 29. PMID 41023216
- [Derived] Ikoma N, Grotz T, Kawakubo H, Kim HI, Matsuda S, Hirata Y, Nakao A, Williams LA, Wang XS, Mendoza T, Wang X, Badgwell BD, Mansfield PF, Hyung WJ, Strong VE, Kitagawa Y. Trans-pacific multicenter collaborative study of minimally invasive proximal versus total gastrectomy for proximal gastric and gastroesophageal junction cancers. BMC Surg. 2023 Sep 1;23(1):262. doi: 10.1186/s12893-023-02163-8. PMID 37653380
- See also: M D Anderson Cancer Center — http://www.mdanderson.org